CLINICAL TRIAL: NCT01042392
Title: Efficacy of Aliskiren Compared to Ramipril in the Treatment of Moderate Systolic Hypertensive Patients
Acronym: ALIAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100AFR01; 2009-011296-80 (EudraCT Number)
Record Dates: First submitted 2010-01-01; First posted 2010-01-05 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Essential Hypertension
Keywords: Moderate systolic hypertension - adults - aliskiren -ramipril
MeSH Terms: conditions — Essential Hypertension | interventions — aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Ramipril (Active Comparator): In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Ramipril 5 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to Ramipril 10 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, part of patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
  Interventions: Drug: Ramipril; Drug: Matching placebo to Aliskiren
- Aliskiren (Experimental): In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Aliskiren 150 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to aliskiren 300 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal ): At visit 4, part of the patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
  Interventions: Drug: Aliskiren; Drug: Matching placebo to Ramipril
- Placebo to Ramipril (Placebo Comparator): In period III (double-blind withdrawal ): At visit 4, part of patients from Ramipril arm received placebo to Ramipril for 1 day. The study ended at visit 5 (48 hours later than visit 4).
  Interventions: Drug: Matching placebo to Ramipril
- Placebo to Aliskiren (Placebo Comparator): In period III (double-blind withdrawal ): At visit 4, part of the patients from Aliskiren arm received placebo to Aliskiren for 1 day. The study ended at visit 5 (48 hours later than visit 4).
  Interventions: Drug: Matching placebo to Aliskiren

INTERVENTIONS:
Drug: Aliskiren — 150 mg Aliskiren as film-coated tablet
  Arms: Aliskiren
Drug: Ramipril — Ramipril 5 mg was given in capsule form.
  Arms: Ramipril
Drug: Matching placebo to Aliskiren — The tablet of matching placebo to aliskiren 150 mg for period I and III. In period II, matching placebo to Aliskiren was given to Ramipril active treatment arm.
  Arms: Placebo to Aliskiren; Ramipril
Drug: Matching placebo to Ramipril — The placebo capsule to ramipril 5 mg for period I and III. In period II, matching placebo to Ramipril was given to Aliskiren active treatment arm.
  Arms: Aliskiren; Placebo to Ramipril

SUMMARY:
This prospective multicenter, double blind study will evaluate the efficacy and safety of aliskiren versus ramipril in patients with moderate systolic essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients > 18 years
* Male or female patients. Female patients must have been either post-menopausal for one year, surgically sterile, or using effective contraceptive methods
* Patients with essential hypertension, previously treated with an antihypertensive single-drug therapy, either uncontrolled or intolerant.
* BP thresholds at visit 1:

  * For patients previously treated and uncontrolled: 140≤ office SBP<180 mmHg
  * For patients previously treated, controlled but intolerant: office SBP≥130 mmHg
* BP thresholds at visit 2 (for all patients):

  * 160≤office SBP<180 mmHg AND
  * 155≤home SBP<175 mmHg (3-day period of home blood pressure monitoring just before randomization)

Exclusion Criteria:

* Women of child-bearing potential not using any effective methods of contraception
* Severe hypertension (office BP ≥ 180/110 mmHg)
* Impossibility to stop abruptly previous antihypertensive treatments at visit 1
* Patients previously untreated or patients treated with two or three antihypertensive medications
* History or evidence of a secondary form of hypertension
* History of hypersensitivity to ACEi or renin inhibitors
* History of heart failure, stroke or coronary heart disease
* Serum potassium ≥ 5.2 mmol/l

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (98):
- France (98):
  - Novartis Investigative Site, Aire Sur Adour
  - Novartis Investigative Site, Amboise
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Anzin
  - Novartis Investigative Site, Bachant
  - Novartis Investigative Site, Bandol
  - Novartis Investigative Site, Bersée
  - Novartis Investigative Site, Bécon-les-Granits
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bouliac
  - Novartis Investigative Site, Bourges
  - Novartis Investigative Site, Briollay
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Carbonne
  - Novartis Investigative Site, Chatillon Sur Colmon
  - Novartis Investigative Site, Château-Gontier
  - Novartis Investigative Site, Châtellerault
  - Novartis Investigative Site, Cherbourg
  - Novartis Investigative Site, Cournonterral
  - Novartis Investigative Site, Croix
  - Novartis Investigative Site, Cugnaux
  - Novartis Investigative Site, Écouflant
  - Novartis Investigative Site, Équeurdreville-Hainneville
  - Novartis Investigative Site, Falaise
  - Novartis Investigative Site, Fondettes
  - Novartis Investigative Site, Guérigny
  - Novartis Investigative Site, Hautmont
  - Novartis Investigative Site, L'Aigle
  - Novartis Investigative Site, La Farlède
  - Novartis Investigative Site, La Riche
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Labarthe-sur-Lèze
  - Novartis Investigative Site, Lambersart
  - Novartis Investigative Site, Laval
  - Novartis Investigative Site, Le Bouscat
  - Novartis Investigative Site, Le Cailar
  - Novartis Investigative Site, Le Fousseret
  - Novartis Investigative Site, Le Pradet
  - Novartis Investigative Site, Les Maguelone
  - Novartis Investigative Site, Luynes
  - Novartis Investigative Site, Marcheprime
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Marsilly
  - Novartis Investigator Site, Marsilly
  - Novartis Investigative Site, Mayenne
  - Novartis Investigative Site, Médis
  - Novartis Investigative Site, Mont-de-Marsan
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Montrevault
  - Novartis Investigative Site, Monts-sur-Guesnes
  - Novartis Investigative Site, Mortagne-sur-Sèvre
  - Novartis Investigative Site, Mourmelon-le-Petit
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nevers
  - Novartis Investigative Site, Nieul-sur-Mer
  - Novartis Investigative Site, Orchies
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Périgny
  - Novartis Investigative Site, Potigny
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Roquevaire
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Avertin
  - Novartis Investigative Site, Saint-Benoît
  - Novartis Investigative Site, Saint-Cyr-sur-Loire
  - Novartis Investigative Site, Saint-Cyr-sur-Mer
  - Novartis Investigative Site, Saint-Georges-dOrques
  - Novartis Investigative Site, Saint-Germain-de-Marencennes
  - Novartis Investigative Site, Saint-Loubès
  - Novartis Investigative Site, Saint-Martin-d'Oney
  - Investigative Site, Saint-Orens-de-Gameville
  - Novartis Investigative Site, Saint-Orens-de-Gameville
  - Novartis Investigative Site, Saint-Rogatien
  - Novartis Investigative Site, Saint-Seurin-de-Cursac
  - Novartis Investigative Site, Saint-Xandre
  - Novartis Investigative Site, Sainte-Marie-de-Ré
  - Novartis Investigative Site, Sanary-sur-Mer
  - Novartis Investigative Site, Savonnières
  - Investigative Site, Scorbé-Clairvaux
  - Novartis Investigative Site, Scorbé-Clairvaux
  - Novartis Investigative Site, Segré
  - Novartis Investigative Site, Seysses
  - Novartis Investigative Site, Sotteville-lès-Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Thun-Saint-Amand
  - Novartis Investigative Site, Tiercé
  - Investigative Site, Toulon
  - Novartis Investigative Site, Toulon
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Trélazé
  - Novartis Investigative Site, Vendôme
  - Novartis Investigative Site, Vereneque
  - Novartis Investigative Site, Verzy
  - Novartis Investigative Site, Vierzon
  - Novartis Investigative Site, Vieux-Condé
  - Novartis Investigative Site, Witry-lès-Reims

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramipril: In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Ramipril 5 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to Ramipril 10 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Placebo to Ramipril: In period III (double-blind withdrawal): At visit 4, part of the patients from Ramipril arm received placebo to Ramipril for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Aliskiren: In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Aliskiren 150 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to aliskiren 300 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, part of patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Placebo to Aliskiren: In period III (double-blind withdrawal): At visit 4, part of patients from Aliskiren arm received placebo for 1 day. The study ended at visit 5 (48 hours later than visit 4).
Period: Period II(Randomized,Double Blinded,8wk)
Arm/Group | Ramipril | Placebo to Ramipril | Aliskiren | Placebo to Aliskiren
Started | 257 | 0 (This arm is used only in Period III.) | 249 | 0 (This arm is used only in Period III.)
Intent to Treat (ITT) | 222 (ITT excluded patients from centers where 90% of BP measurements were rounded to 5 or 0) | 0 | 222 | 0
Completed | 247 | 0 | 241 | 0
Not Completed | 10 | 0 | 8 | 0
Not completed — Adverse Event | 6 | 0 | 5 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Administrative problems | 2 | 0 | 0 | 0
Period: Period III (Unblinded,Controlled, 1 Day)
Arm/Group | Ramipril | Placebo to Ramipril | Aliskiren | Placebo to Aliskiren
Started | 129 | 118 | 119 | 122
Per Protocol Missed-dose (PPMD) | 98 (PPMD excluded patients violated protocol instructions for period 3 (duration and treatment intake)) | 73 | 93 | 82
Completed | 127 | 117 | 115 | 121
Not Completed | 2 | 1 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Administrative problems | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ramipril: In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Ramipril 5 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to Ramipril 10 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, patients received placebo or the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Aliskiren: In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Aliskiren 150 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to aliskiren 300 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, patients received placebo or the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Total: Total of all reporting groups
Arm/Group | Ramipril | Aliskiren | Total
Number analyzed (Participants) | 257 | 249 | 506
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.6) | 61.0 (11.4) | 60.4 (11.5)
Age, Customized [Number; unit: Participants]
  < 50 years | 56 | 39 | 95
  50 - 64 years | 119 | 115 | 234
  65 - 74 years | 56 | 64 | 120
  >= 75 years | 26 | 31 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 133 | 275
  Male | 115 | 116 | 231

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: The arm in which the highest sitting systolic blood pressure (SBP) was found at study entry was used for all subsequent readings. At each study visit, after leaving the patient to rest 5 minutes in a sitting position, the blood pressure (BP) was measured three times with an oscillometric device. The measurements were performed at 1-2 minute intervals. The mean BP was calculated from the 3 readings. The analysis of covariance included treatment factor and baseline mean sitting SBP as covariable.
Time Frame: Baseline to 8 weeks
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 213 | 213
mmHg | -18.80 (0.92) | -20.78 (0.92)

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: The arm in which the highest sitting systolic blood pressure (SBP) was found at study entry was used for all subsequent readings. At each study visit, after leaving the patient to rest 5 minutes in a sitting position, the blood pressure (BP) was measured three times with an oscillometric device. The measurements were performed at 1-2 minute intervals. The mean BP was calculated from the 3 readings. The analysis of variance included treatment factor and baseline value of mean sitting DBP as covariable.
Time Frame: Baseline to 8 weeks
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5. Patients with observation at both time points were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 213 | 213
mmHg | -5.23 (0.60) | -6.39 (0.60)

3. Secondary Outcome: Percentage of Patients With Controlled Blood Pressure
Description: The arm in which the highest sitting systolic blood pressure (SBP) was found at study entry was used for all subsequent readings. At each study visit, after leaving the patient to rest 5 minutes in a sitting position, the blood pressure (BP) was measured three times with an oscillometric device. The measurements were performed at 1-2 minute intervals. The mean BP was calculated from the 3 readings.
  Controlled blood pressure (BP) is defined as mean office systolic BP/ diastolic BP < 140/90 mmHg.
Time Frame: At 4 and 8 weeks
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5. Patients with observation at each time point were included in this analysis.
Measure: Number; unit: Percentage
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 222 | 222
Percentage
  At week 4 (N= 218, 217) | 36.7 | 40.1
  At week 8 (N= 213, 213) | 26.8 | 32.4

4. Secondary Outcome: Number of the Participants With More Than 55 mmHg Difference Between the Mean SBP Measured at the Morning Surge and the Mean Minimal SBP Measured During the Night
Description: Ambulatory blood pressure measurement (ABPM) over 24 hours was performed for all patients on the day before visit 4, the device attached to the ambulatory blood pressure non-dominant arm of the patient. The BP morning surge was defined as the average of the measurements taken during the first 2 hours after waking the patient. The minimal night blood pressure was defined as the average of the two lowest BP measures (the lowest hourly average) recorded during night time.
Time Frame: After 8 weeks
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5. Patients with ABPM to evaluate the occurrence or absence of a morning peak were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 114 | 112
Participants | 3 | 9

5. Secondary Outcome: Change in msSBP and msDBP From Visit 2 (Baseline) to Visit 3 (at 4 Weeks)
Description: The arm in which the highest sitting systolic blood pressure (SBP) was found at study entry was used for all subsequent readings. At each study visit, after leaving the patient to rest 5 minutes in a sitting position, the blood pressure (BP) was measured three times with an oscillometric device. The measurements were performed at 1-2 minute intervals. The mean BP was calculated from the 3 readings. The analysis of covariance included treatment factor and baseline mean sitting SBP and mean sitting DBP as covariables.
Time Frame: Baseline to 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 218 | 217
mmHg
  Change in msSBP | -19.42 (0.92) | -19.75 (0.92)
  Change in msDBP | -5.37 (0.56) | -5.60 (0.56)

6. Secondary Outcome: Difference Between the Maximal and the Minimal Mean-hour SPB Measured Between 1 and 8 am at Week 8
Description: Ambulatory blood pressure measurement (ABPM) over 24 hours was performed for all patients on the eve of visit 4 (week 8), the device attached to the ambulatory blood pressure non-dominant arm of the patient. The difference between mean-hour maximum SBP mean-hour minimum SBP between 1 am and 8 am was measured.
Time Frame: At week 8
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5. Patients with ABPM measurements over 24 hours were included in this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 175 | 186
mmHg | 33.6 (14.04) | 35.5 (15.05)

7. Secondary Outcome: Change in Mean Sitting DBP and SBP in Specified Sub-groups From Visit 2 (Baseline) to Visit 4 (at 8 Weeks)
Description: The sub-groups were: "Riser" = patients with >= 55 mmHg difference between the mean SPB measured at the morning surge and the mean minimal SBP measured during the night. The "Non-risers" in whom the difference is <55 mmHg. Patients called "dippers" in whom there was a decrease in average nocturnal SBP ≥ 10% compared with average daytime SBP, in contrast to patients "non-dippers " in whom this difference was <10%.
Time Frame: Baseline to 8 weeks
Population: Intent to treat population included all randomized patients who had received at least one dose of study drug. It also excluded all those patients from centers that reported more than 90% of BP measurements rounded to 0 or 5. Patients with observation at different categories were included in this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 222 | 222
mmHg
  Change in msSBP: Risers (n= 3, 9) | -19.7 (6.11) | -16.9 (10.52)
  Change in msSBP: Non-risers (n=109, 103) | -19.2 (13.99) | -20.5 (14.49)
  Change in msSBP: Dippers (n= 80, 94) | -18.1 (11.86) | -19.8 (12.05)
  Change in msSBP: Non-dippers (n= 93, 92) | -19.2 (14.93) | -21.1 (15.06)
  Change in msDBP: Risers (n= 3, 9) | -7.3 (10.60) | -6.6 (9.11)
  Change in msDBP: Non-risers(n=109, 103) | -4.2 (9.51) | -5.7 (9.61)
  Change in msDBP: Dippers (n= 80, 94) | -5.5 (9.63) | -6.3 (9.81)
  Change in msDBP: Non-dippers (n= 93, 92) | -5.3 (9.59) | -6.5 (9.56)

8. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP) From Last Active Dose Taken to After a One-day Missed-dose
Description: The change in blood pressure was measured between visit 4 (end of the period of double-blind active treatment which was at week 8) and visit 5 (48 hours after the last active dose taken) in the group of patients who received aliskiren or placebo and those who received ramipril or placebo. The analysis of covariance included treatment factor and baseline mean sitting SBP and mean sitting DBP as covariables.
Time Frame: From 8 weeks to 48 hours after week 8
Population: Per-protocol missed dose population included all per protocol population patients who had received the study treatment for period 3 according to the protocol (duration of period 3 and treatment intake). Patients with observation at both time points were included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Ramipril | Placebo to Ramipril | Aliskiren | Placebo to Aliskiren
Number analyzed (Participants) | 95 | 73 | 88 | 81
mmHg
  Change in msSBP | -0.50 (1.05) | -1.28 (1.10) | 0.52 (1.06) | 3.27 (1.10)
  Change in msDBP | 0.76 (0.69) | 0.32 (0.79) | -0.40 (0.78) | 0.97 (0.81)

9. Secondary Outcome: Number Patients Reported With Adverse Events (AEs), Serious Adverse Events (SAE) and Death (Period II and Period III)
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 8 weeks + 1 day
Population: All randomized patients except one patient from Aliskiren arm who was lost to follow up after visit 2.
Measure: Number; unit: Participants
Arm/Group | Ramipril | Aliskiren
Number analyzed (Participants) | 257 | 248
Participants
  Patients with at least 1 AE | 55 | 43
  Patients with at least 1 SAE | 3 | 1
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks of period II + 1 day of Period III
Description: The adverse events and serious adverse events are reported on randomized population except one patient who lost to follow up after visit 2.
Groups:
- Ramipril (Period II and III): In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Ramipril 5 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to Ramipril 10 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Placebo to Ramipril (Period III): In period III (double-blind withdrawal): At visit 4, part of the patients from Ramipril arm received placebo to Ramipril for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Aliskiren (Period II and III): In period I (washout and single-blind): from visit 1 to visit 2, 2 weeks placebo run-in.
  In period II (double-blind treatment, randomized): Aliskiren 150 mg for 4 weeks (visit 2 - visit 3). At visit 3, medications had to be titrated to aliskiren 300 mg only if BP remained ≥ 140/90 mmHg. Double blind treatment had to be continued for another 4-week period until visit 4.
  In period III (double-blind withdrawal): At visit 4, part of patients received the active treatment for 1 day. The study ended at visit 5 (48 hours later than visit 4).
- Placebo to Aliskiren (Period III): In period III (double-blind withdrawal): At visit 4, part of patients from Aliskiren arm received placebo for 1 day. The study ended at visit 5 (48 hours later than visit 4).
Arm/Group | Ramipril (Period II and III) | Placebo to Ramipril (Period III) | Aliskiren (Period II and III) | Placebo to Aliskiren (Period III)
Serious Adverse Events (participants affected / at risk) | 3/257 | 0/118 | 1/248 | 0/122
Other Adverse Events (participants affected / at risk) | 0/257 | 0/118 | 0/248 | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramipril (Period II and III) (N=257) | Placebo to Ramipril (Period III) (N=118) | Aliskiren (Period II and III) (N=248) | Placebo to Aliskiren (Period III) (N=122)
normochromic normocytic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
spine metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
liver metastatis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
asthenia (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.